CLINICAL TRIAL: NCT01478165
Title: Comparative Study of TIVA(Total Intravenous Anesthesia) and TIVA Plus Palonosetron in Preventing PONV(Postoperative Nausea and Vomiting)
Brief Title: Comparison of TIVA (Total Intravenous Anesthesia) and TIVA Plus Palonosetron in Preventing Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Soo Kyoung Park, Clnical professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OC11MISI0090
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Palonosetron; PONV(postoperative nausea and vomiting); TIVA(Total intravenous anesthesia)
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tiva group (Group T) (Placebo Comparator)
  Interventions: Drug: Total intravenous anesthesia
- TIVA plus palonosetron group (Group T+P) (Active Comparator)
  Interventions: Drug: Total intravenous anesthesia plus palonosetron

INTERVENTIONS:
Drug: Total intravenous anesthesia — Total intravenous anesthesia plus normal saline 1.5 ml immediately before induction of anesthesia
  Arms: Tiva group (Group T)
Drug: Total intravenous anesthesia plus palonosetron — Total intravenous anesthesia plus palonosetron 0.075 mg(1.5 ml)immediately before induction of anesthesia
  Arms: TIVA plus palonosetron group (Group T+P)

SUMMARY:
A total intravenous anesthesia (TIVA) is a useful anesthetic technique that reduces the incidence of postoperative nausea and vomiting (PONV).

Investigator hypothesized the incidence of PONV can be further reduced when palonosetron is added to TIVA.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1 or 2
* Elective gynaecological laparoscopic surgery of ≥ 1h duration

Exclusion Criteria:

* Anti-emetics, steroids, or psychoactive medications within 24 h of study initiation
* Vomiting or retching in the 24 h preceding surgery
* Cancer chemotherapy within 4 weeks or emetogenic radiotherapy within 8 weeks before study entry
* Ongoing vomiting from gastrointestinal disease

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting | For 24 hours after surgery

SECONDARY OUTCOMES:
Severity of nausea | For 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Soo Kyoung Park, Principal Investigator — Incheon St.Mary's Hospital
Locations (1):
- Incheon St. Mary's hospital, Incheon, South Korea